CLINICAL TRIAL: NCT01291667
Title: A Phase III Randomized Study for HER2-Overexpressed Metastatic Breast Cancer Patients Treated by Trastuzumab( Cipterbin®) Plus vinorelbinE Simultaneously or Sequencely
Brief Title: Study for HER2-Overexpressed MBC Patients Treated by Cipterbin® Plus vinorelbinE
Acronym: HOPES
Status: Completed | Type: Observational
Sponsor: Shanghai CP Guojian Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Zefei Jiang, Hospital Affiliated to Academy Military Medical Science
Other Study IDs: HOPES
Record Dates: First submitted 2011-02-06; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-02

CONDITIONS: Progress-free Survival; Overall Response Rate; Adverse Events

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Breast cancer is the most common malignant disease and the most frequent causes of cancer mortality in females worldwide. The situation is same as the world in China. Trastuzumab has been proved valuable treatment for HER2-positive breast cancer patients. Cipterbin® is developing by Shanghai CP Guojian Pharmaceutical Co.Ltd.Now we carried on the phase III trial in order to prove Cipterbin® 's efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* signed ICF
* pathologic diagnosis breast cancer
* HER2+ status defined as IHC3+ Staining or in situ hybridization positive at least 1 measurable lesion as per RECIST criteria age from 18y to 70y KPS>=70

Exclusion Criteria:

* More than three prior chemotherapy lines for advanced disease LVEF<50%
* prior exposure vinorebine for breast cancer
* prior exposure Trastuzumab for breast cancer
* uncontrolled brain metastasis
* breastfeeding or pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive metastatic breast cancer patients
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2009-05

PRIMARY OUTCOMES:
progress-free survival

SECONDARY OUTCOMES:
overall response rate,safety